CLINICAL TRIAL: NCT05535322
Title: Real-world Evaluation of GLP-1 Receptor Agonists (GLP-1RA) on Efficacy and Persistence, Adherence and Therapeutic Inertia Among Type 2 Diabetes Adults With Obesity in the Department of Health of Valencia Clínico-Malvarrosa
Brief Title: Real-world Evaluation of GLP-1 Receptor Agonists (GLP-1RA) on Efficacy and Persistence, Adherence and Therapeutic Inertia Among Type 2 Diabetes Adults With Obesity
Status: Completed | Type: Observational
Sponsor: Ana Palanca (Other)
Responsible Party: Sponsor-Investigator, Ana Palanca, Clinical Research Coordinator, Fundación para la Investigación del Hospital Clínico de Valencia
Organization: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Other Study IDs: GLP-1RA in T2D
Record Dates: First submitted 2022-03-07; First posted 2022-09-10 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GLP-1RA: All GLP-1RA users: all T2D adults treated with GLP-1RA or initiating a GLP-1RA during the study period
  Interventions: Drug: GLP-1RA
- SGLT2i: SGLT2 inhibitors users with no GLP-1RA prescription: all T2D adults treated with SGLT2i or initiating treatment with SGLT2i during the study period and who were not treated with a GLP-1RA
  Interventions: Drug: SGLT2i
- Insulin: Insulin users with no GLP-1RA and/or SGLT2i prescriptions: all T2D adults treated with insulin or initiating insulin treatment during the study period and who were not treated with GLP-1RA/SGLT2i
  Interventions: Drug: Insulin
- Miscellany: Other glucose-lowering agents users: all T2D adults who were not treated with GLP-1RA and/or SGLT2i and/or insulin during the study period.
  Interventions: Drug: Miscellany

INTERVENTIONS:
Drug: GLP-1RA — All T2D adults treated with Glucagon-like peptide-1 receptor agonists (GLP-1RA) or initiating a GLP-1RA during the study period
  Groups: GLP-1RA
Drug: SGLT2i — SGLT2 inhibitors users with no GLP-1RA prescription: all T2D adults treated with Sodium/glucose cotransporter-2 inhibitors (SGLT2i) or initiating treatment with SGLT2i during the study period and who were not treated with a GLP-1RA
  Groups: SGLT2i
Drug: Insulin — Insulin users with no GLP-1RA and/or SGLT2i prescriptions: all T2D adults treated with insulin or initiating insulin treatment during the study period and who were not treated with GLP-1RA/SGLT2i
  Groups: Insulin
Drug: Miscellany — Other glucose-lowering agents users: all T2D adults who were not treated with GLP-1RA and/or SGLT2i and/or insulin during the study period and who were treated with other glucose-lowering agents during the study period
  Groups: Miscellany

SUMMARY:
Type 2 diabetes (T2D) is a progressive chronic condition associated with a high morbi-mortality that has a considerable impact on healthcare resources.

Glucagon-like peptide-1 receptor agonists (GLP-1RA) are incretin mimetics that have been shown to improve glycemic control with a low associated risk of hypoglycemia. Additionally, previous studies have linked the use of GLP-1RA with a reduction in the risk of cardiovascular events and kidney disease progression. Despite these positive results, GLP1-RA´s prescription, following the failure of treatment with metformin monotherapy or dual therapy, remains low in Spain compared to other countries in our milieu. Furthermore, the use of this therapeutic class is not homogeneous across the different autonomous communities in Spain, and, no objective justification for these differences seems to exist. Consequently, there is a need to understand which are the benefits associated with the use of GLP-1RA, versus intensification with other oral agents, in real-life conditions.

In this study, the impact of the use of GLP-1RA on clinical outcomes such as all-cause mortality, cardiovascular and renal outcomes as well as severe hypoglycemia will be evaluated based on the analysis of longitudinal databases that collect the variables of interest generated in a real-life scenario. In addition, both persistence and adherence to treatment in patients treated with GLP-1RA and its impact on the clinical outcomes of interest will be studied. Finally, therapeutic inertia will be analyzed.

All these data will contribute to generating cost-effective strategies aimed at improving health outcomes among T2D patients in our setting, reinforcing persistence and adherence to the prescribed treatment, and reducing therapeutic inertia in this group of patients.

Since the use of GLP-1RA versus intensification with other oral agents has been associated with better glycemic control, and, when compared to intensification with basal insulin, with a lower incidence of severe hypoglycemia, we hypothesized that T2D adults treated with GLP-1RA would present a lower incidence of cardiovascular and renal outcomes and fewer hospitalizations due to severe hypoglycemia events as well as a decreased all-cause mortality. On the other hand, patients on GLP-1RA who would present greater persistence and adherence to treatment should experience fewer cardiovascular and renal outcomes and lower mortality compared to those with less persistence and adherence. Finally, it is possible that the type of GLP-1RA and the mode of administration, weekly versus daily, may influence adherence, persistence and therapeutic inertia in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults with type 2 diabetes
* Individuals with at least a 6-month prescription

Exclusion Criteria:

* Individuals below 18
* Individuals with less than a 6-month prescription

Ages: 18 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All identified adults with type 2 diabetes registered in the Population Information System (SIP) of the Valencian Community and corresponding to the Valencia Clínico-La Malvarrosa Health Department who were diagnosed before the end of the study period were included. Type 2 diabetes (T2D) diagnosis was defined according to the International Classification of Diseases, Ninth and Tenth Revisions, Clinical Modification (ICD-9-CM, ICD-10-CM) codes.
  To exclude temporary treatment effects due to short-term use of the antidiabetic treatments, only individuals in the study groups with at least a 6-month prescription were included in the analyses.
Sampling Method: Non-Probability Sample
Enrollment: 26944 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Major acute cardiovascular events | From inclusion in the study, starting from 01/01/2014, until the event or the end of the study, on 31/12/2019, whichever came first.
  In this work, this composite includes patients suffering from non-fatal acute myocardial infarction (AMI) and non-fatal stroke, transient ischemic attack (TIA), all-cause death, and, heart failure events occurring during the study period (from inclusion in the study until the event or the end of the study period, whichever came first).

SECONDARY OUTCOMES:
Major acute cardiovascular events without heart failure | From inclusion in the study, starting from 01/01/2014, until the event or the end of the study, on 31/12/2019, whichever came first.
  In this work, this composite includes patients suffering from non-fatal acute myocardial infarction (AMI) and non-fatal stroke, transient ischemic attack (TIA) and all-cause death occurring during the study period (from inclusion in the study until the event or the end of the study period, whichever came first).
AMI | From inclusion in the study, starting from 01/01/2014, until the event or the end of the study, on 31/12/2019, whichever came first.
  Acute myocardial infarction events occurring during the study follow-up (from inclusion in the study until the event or the end of the study period, whichever came first.
Stroke | From inclusion in the study, starting from 01/01/2014, until the event or the end of the study, on 31/12/2019, whichever came first.
  Stroke events occurring during the study follow-up (from inclusion in the study until the event or the end of the study period, whichever came first.
Heart Failure | Through study completion (from inclusion in the study until the event or the end of the study period, whichever came first)
  Heart failure hospitalization occurring during the study follow-up (from inclusion in the study until the event or the end of the study period, whichever came first.
all-cause death | From inclusion in the study, starting from 01/01/2014, until the event or the end of the study, on 31/12/2019, whichever came first.
  Death from all causes occurring during the study follow-up (from inclusion in the study until the event or the end of the study period, whichever came first.
Renal progression | From inclusion in the study, starting from 01/01/2014, until the event or the end of the study, on 31/12/2019, whichever came first.
  Sustained 40% reduction in eGFR occurring during the study follow-up (from inclusion in the study until the event or the end of the study period, whichever came first.
atrial fibrillation | From inclusion in the study, starting from 01/01/2014, until the event or the end of the study, on 31/12/2019, whichever came first.
  Events of atrial fibrillation episodes occurring during the study follow-up (from inclusion in the study until the event or the end of the study period, whichever came first.
Hypoglycemia | From inclusion in the study, starting from 01/01/2014, until the event or the end of the study, on 31/12/2019, whichever came first.
  Severe hypoglycemia requiring hospitalization occurring during the study follow-up (from inclusion in the study until the event or the end of the study period, whichever came first.
Persistence | From inclusion in the study, starting from 01/01/2014, until the end of the study, on 31/12/2019.
  Persistence on treatment was defined as the percentage of patients continuing treatment from the start of the study period or since the first prescription during the study period until evidence of discontinuation or the end of the study period.
Adherence | From inclusion in the study, starting from 01/01/2014, until the end of the study, on 31/12/2019.
  Treatment adherence was defined as the proportion of days covered (days in which an individual had access to the medication) from the start of the study period or since the first prescription during the study period until treatment discontinuation
Therapeutic inertia | From inclusion in the study, starting from 01/01/2014, until the end of the study, on 31/12/2019.
  Therapeutic inertia was defined as non-intensification of treatment once started despite HbA1c ≥7.5% during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- INCLIVA, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blonde L, Raccah D, Lew E, Meyers J, Nikonova E, Ajmera M, Davis KL, Bertolini M, Guerci B. Treatment Intensification in Type 2 Diabetes: A Real-World Study of 2-OAD Regimens, GLP-1 RAs, or Basal Insulin. Diabetes Ther. 2018 Jun;9(3):1169-1184. doi: 10.1007/s13300-018-0429-x. Epub 2018 Apr 19. PMID 29675797
- [Background] Carls GS, Tuttle E, Tan RD, Huynh J, Yee J, Edelman SV, Polonsky WH. Understanding the Gap Between Efficacy in Randomized Controlled Trials and Effectiveness in Real-World Use of GLP-1 RA and DPP-4 Therapies in Patients With Type 2 Diabetes. Diabetes Care. 2017 Nov;40(11):1469-1478. doi: 10.2337/dc16-2725. Epub 2017 Aug 11. PMID 28801475
- [Background] Chatterjee S, Davies MJ, Khunti K. What have we learnt from "real world" data, observational studies and meta-analyses. Diabetes Obes Metab. 2018 Feb;20 Suppl 1:47-58. doi: 10.1111/dom.13178. PMID 29364585
- [Background] Conget I, Mauricio D, Ortega R, Detournay B; CHADIG Study investigators. Characteristics of patients with type 2 diabetes mellitus newly treated with GLP-1 receptor agonists (CHADIG Study): a cross-sectional multicentre study in Spain. BMJ Open. 2016 Jul 26;6(7):e010197. doi: 10.1136/bmjopen-2015-010197. PMID 27466235
- [Background] Divino V, Boye KS, Lebrec J, DeKoven M, Norrbacka K. GLP-1 RA Treatment and Dosing Patterns Among Type 2 Diabetes Patients in Six Countries: A Retrospective Analysis of Pharmacy Claims Data. Diabetes Ther. 2019 Jun;10(3):1067-1088. doi: 10.1007/s13300-019-0615-5. Epub 2019 Apr 26. PMID 31028689
- [Background] Divino V, DeKoven M, Khan FA, Boye KS, Sapin H, Norrbacka K. GLP-1 RA Treatment Patterns Among Type 2 Diabetes Patients in Five European Countries. Diabetes Ther. 2017 Feb;8(1):115-128. doi: 10.1007/s13300-016-0224-5. Epub 2017 Jan 9. PMID 28070733
- [Background] Fadini GP, Frison V, Rigato M, Morieri ML, Simioni N, Tadiotto F, D'Ambrosio M, Paccagnella A, Lapolla A, Avogaro A. Trend 2010-2018 in the clinical use of GLP-1 receptor agonists for the treatment of type 2 diabetes in routine clinical practice: an observational study from Northeast Italy. Acta Diabetol. 2020 Mar;57(3):367-375. doi: 10.1007/s00592-019-01445-z. Epub 2019 Oct 31. PMID 31673896
- [Background] Fu AZ, Qiu Y, Davies MJ, Radican L, Engel SS. Treatment intensification in patients with type 2 diabetes who failed metformin monotherapy. Diabetes Obes Metab. 2011 Aug;13(8):765-9. doi: 10.1111/j.1463-1326.2011.01405.x. PMID 21457427
- [Background] Gaede P, Oellgaard J, Carstensen B, Rossing P, Lund-Andersen H, Parving HH, Pedersen O. Years of life gained by multifactorial intervention in patients with type 2 diabetes mellitus and microalbuminuria: 21 years follow-up on the Steno-2 randomised trial. Diabetologia. 2016 Nov;59(11):2298-2307. doi: 10.1007/s00125-016-4065-6. Epub 2016 Aug 16. PMID 27531506
- [Background] Guerci B, Charbonnel B, Gourdy P, Hadjadj S, Hanaire H, Marre M, Verges B. Efficacy and adherence of glucagon-like peptide-1 receptor agonist treatment in patients with type 2 diabetes mellitus in real-life settings. Diabetes Metab. 2019 Dec;45(6):528-535. doi: 10.1016/j.diabet.2019.01.006. Epub 2019 Jan 21. PMID 30677504
- [Background] Hernandez AF, Green JB, Janmohamed S, D'Agostino RB Sr, Granger CB, Jones NP, Leiter LA, Rosenberg AE, Sigmon KN, Somerville MC, Thorpe KM, McMurray JJV, Del Prato S; Harmony Outcomes committees and investigators. Albiglutide and cardiovascular outcomes in patients with type 2 diabetes and cardiovascular disease (Harmony Outcomes): a double-blind, randomised placebo-controlled trial. Lancet. 2018 Oct 27;392(10157):1519-1529. doi: 10.1016/S0140-6736(18)32261-X. Epub 2018 Oct 2. PMID 30291013
- [Background] Kristensen SL, Rorth R, Jhund PS, Docherty KF, Sattar N, Preiss D, Kober L, Petrie MC, McMurray JJV. Cardiovascular, mortality, and kidney outcomes with GLP-1 receptor agonists in patients with type 2 diabetes: a systematic review and meta-analysis of cardiovascular outcome trials. Lancet Diabetes Endocrinol. 2019 Oct;7(10):776-785. doi: 10.1016/S2213-8587(19)30249-9. Epub 2019 Aug 14. PMID 31422062
- [Background] Lin J, Lingohr-Smith M, Fan T. Real-world medication persistence and outcomes associated with basal insulin and glucagon-like peptide 1 receptor agonist free-dose combination therapy in patients with type 2 diabetes in the US. Clinicoecon Outcomes Res. 2016 Dec 22;9:19-29. doi: 10.2147/CEOR.S117200. eCollection 2017. PMID 28053550
- [Background] Leiter LA, Bain SC, Bhatt DL, Buse JB, Mazer CD, Pratley RE, Rasmussen S, Ripa MS, Vrazic H, Verma S. The effect of glucagon-like peptide-1 receptor agonists liraglutide and semaglutide on cardiovascular and renal outcomes across baseline blood pressure categories: Analysis of the LEADER and SUSTAIN 6 trials. Diabetes Obes Metab. 2020 Sep;22(9):1690-1695. doi: 10.1111/dom.14079. Epub 2020 Jun 3. PMID 32372454
- [Background] Khunti K, Gomes MB, Pocock S, Shestakova MV, Pintat S, Fenici P, Hammar N, Medina J. Therapeutic inertia in the treatment of hyperglycaemia in patients with type 2 diabetes: A systematic review. Diabetes Obes Metab. 2018 Feb;20(2):427-437. doi: 10.1111/dom.13088. Epub 2017 Oct 1. PMID 28834075
- [Background] Pasternak B, Wintzell V, Eliasson B, Svensson AM, Franzen S, Gudbjornsdottir S, Hveem K, Jonasson C, Melbye M, Svanstrom H, Ueda P. Use of Glucagon-Like Peptide 1 Receptor Agonists and Risk of Serious Renal Events: Scandinavian Cohort Study. Diabetes Care. 2020 Jun;43(6):1326-1335. doi: 10.2337/dc19-2088. Epub 2020 Apr 15. PMID 32295809
- [Background] Pineda ED, Liao IC, Godley PJ, Michel JB, Rascati KL. Cardiovascular Outcomes Among Patients with Type 2 Diabetes Newly Initiated on Sodium-Glucose Cotransporter-2 Inhibitors, Glucagon-Like Peptide-1 Receptor Agonists, and Other Antidiabetic Medications. J Manag Care Spec Pharm. 2020 May;26(5):610-618. doi: 10.18553/jmcp.2020.26.5.610. PMID 32347181
- [Derived] Palanca A, Ampudia-Blasco FJ, Calderon JM, Sauri I, Martinez-Hervas S, Trillo JL, Redon J, Real JT. Real-World Evaluation of GLP-1 Receptor Agonist Therapy Persistence, Adherence and Therapeutic Inertia Among Obese Adults with Type 2 Diabetes. Diabetes Ther. 2023 Apr;14(4):723-736. doi: 10.1007/s13300-023-01382-9. Epub 2023 Feb 27. PMID 36847952